CLINICAL TRIAL: NCT01685268
Title: A Study of HSP90 Inhibitor AT13387 Alone or in Combination With Abiraterone Acetate in the Treatment of Castration-Resistant Prostate Cancer (CRPC) no Longer Responding to Abiraterone
Brief Title: A Study of HSP90 Inhibitor AT13387 Alone or in Combination With Abiraterone Acetate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AT13387-04
Record Dates: First submitted 2012-08-31; First posted 2012-09-14 (Estimated); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone; Abiraterone Acetate; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A, Regimen 1 (Experimental): AT13387 given as a 1-hr IV infusion at a starting dose of 220 mg/m2 once weekly for 3 weeks in a 4-week cycle, in combination with abiraterone acetate 1000 mg by mouth (PO) daily (QD) and prednisone or prednisolone 5 mg PO twice daily.
  Interventions: Drug: AT13387; Drug: abiraterone acetate; Drug: Prednisone
- Part A, Regimen 2 (Experimental): At13387 administered as a 1-hr IV infusion at a starting dose of 120 mg/m2 on Day 1 and Day 2 weekly for 3 weeks in a 4-week cycle, in combination with abiraterone acetate 1000 mg by mouth (PO) daily (QD) and prednisone or prednisolone 5 mg PO twice daily.
  Interventions: Drug: AT13387; Drug: abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: AT13387 — Regimen 1: AT13387, given as 1-hr intravenous infusion at starting dose of 220 mg/m2 once weekly for 3 weeks in a 4-week cycle. Regimen 2: AT13387, given as 1-hr IV infusion at starting dose of 120 mg/m2 on Day 1 and Day 2 weekly for 3 weeks in a 4-week cycle.
  Other Names: onalespib
Drug: abiraterone acetate — 1000 mg PO daily.
Drug: Prednisone — 5 mg PO twice daily.
  Other Names: prednisolone

SUMMARY:
A 2-part, Phase 1-2, open-label, parallel group, randomized study in patients with Castration-Resistant Prostate Cancer (CRPC) who are no longer responding to treatment with abiraterone and steroids. In Part A (Phase 1), patients will continue to receive the same doses of abiraterone and steroids they were receiving prior to study entry and will be randomized to receive 1 of 2 different treatment regimens of AT13387 in combination with abiraterone. Once the best regimen is established in Part A, based on safety and antitumor activity, patients will be randomized to the selected treatment regimen and dose of AT13387 in combination with abiraterone or AT13387 alone in Part B (Phase 2).

ELIGIBILITY:
Inclusion:

1. Must have prostate cancer
2. Have received prior castration by orchiectomy and/or hormone therapy
3. Males >18 years of age
4. Normal activity level for self care
5. Have been receiving abiraterone therapy with a steroid for ≥1 month
6. Have disease progression on abiraterone as defined by either PSA progression, radiographic or bone progression
7. Have adequate bone marrow, liver and kidney function
8. Must be willing to provide pre-existing tumor samples, if this material exists. If pre-existing samples are not available, a sample must be obtained during screening
9. Must be willing and able to provide written informed consent and comply with the protocol and study procedures

Exclusion:

1. Prior anti-cancer treatment with any Heat Shock Protein 90 (HSP90) inhibitor or histone deacetylase (HDAC) inhibitor compound
2. Have received chemotherapy within 4 weeks prior to receiving study drug
3. Prior prostate surgery or radiotherapy within 4 weeks from the first dose of study drug
4. Hypersensitivity to AT13387 or other components of the drug product
5. Treatment with any investigational drug within 4 weeks prior to the first dose of study drug
6. Severe systemic diseases or active uncontrolled infections
7. Presence of a life-threatening illness, medical condition, organ system dysfunction, or other factors
8. Abnormal heart function
9. Other cancer except for adequately treated basal cell or squamous cell carcinoma of the skin, or superficial bladder cancer, or other cancer from which the subject has been disease-free for at least 3 years;
10. No known brain or CNS involvement
11. Unable to receive corticosteroids or history of pituitary or adrenal dysfunction
12. Known history of human immunodeficiency virus (HIV) or seropositive test for hepatitis C virus or hepatitis B virus

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and tolerability of the combination of AT13387 and abiraterone and to select the most promising treatment regimen in CRPC patients who are no longer responding to treatment with abiraterone alone. | 12 months
  * Number of patients with adverse events
  * Change in prostate specific antigen measurement and circulating tumor cell count every 4 weeks
  * Change in tumor measurements by RECIST 1.1 every 12 weeks
Part B: Compare the antitumor activity (response rate per the Prostate Cancer Working Group 2 [PCWG2]) between single-agent AT13387 and combination of AT13387 plus abiraterone in patients who are no longer responding to treatment with abiraterone alone. | 12 months
  * Change in prostate specific antigen measurement and circulating tumor cell count every 4 weeks
  * Change in tumor measurements by RECIST 1.1 every 12 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of combination treatment of AT13387 and abiraterone. | 24 months
  * Area under the plasma concentration versus time curve (AUC) of AT13387 and abiraterone alone and in combination by Week 4
  * Maximum concentration (Cmax) of AT13387 and abiraterone alone and in combination by Week 4
Pharmacodynamics of combination treatment of AT13387 and abiraterone. | 24 months
  CTC enumeration and characterization every 4 weeks.
Progression free survival | 24 months
  Assessment of progression free survival as measured by weeks
Overall survival | 24 months
  Overall survival as measured in weeks

CONTACTS AND LOCATIONS:
Locations (32):
- United States (20):
  - University of California, Los Angeles Institute of Urologic Oncology, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Fort Myers, Fort Myers, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Clinical Research Alliance, Inc., Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The West Clinic, Memphis, Tennessee
  - Northwest Medical Specialists, PLLC, Tacoma, Washington
- Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec, Canada
- Centro Integral Oncologico Clara Campal, Madrid, Spain
- United Kingdom (10):
  - Brighton & Sussex University Hospitals NHS Trust, Brighton
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Velindre Cancer Center, Cardiff
  - University of Surrey, Guildford
  - Charing Cross Hospital, London
  - Royal Marsden Foundation Trust Instute of Cancer Researrch, London
  - The Christie Hospital NHS Trust, Manchester
  - Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Nottingham University Hospitals, Nottingham
  - University Hospital Southampton, Southampton